CLINICAL TRIAL: NCT06567574
Title: Stanford Study of the Validation of the Pre-Interventional Preventive Risk Assessment (PIPRA) Tool In The At-Risk Orthopedic Surgery Population
Brief Title: Stanford PIPRA Validation Study in an Elderly Orthopedic Population
Acronym: PIPRA-ORTHO
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jose R Maldonado, MD, Professor of Medicine and Psychiatry, Stanford University
Other Study IDs: IRB-73341
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Delirium; Postoperative Delirium; Cognitive Impairment
Keywords: Artificial Intelligence; Delirium Risk Factors; Delirium; Postoperative Delirium; Cognitive Impairment
MeSH Terms: conditions — Delirium; Emergence Delirium; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the accuracy of an AI-based tool in the prediction of postoperative delirium (POD), in a population at moderately high risk of developing this syndrome (i.e., elderly orthopedic subjects). The population to be studied has already been enrolled in a parallel study regarding the likelihood of developing delirium, its relationship to the type of anesthetic, and the relationship between anesthetic type, development of delirium and risk for post-operative cognitive impairment (including risk for dementia) (Protocol ID#55169 [David Drover-Principal investigator; José Maldonado-Co-investigator]).

DETAILED DESCRIPTION:
Study investigators would like to determine the real-life accuracy of a new tool developed for the prediction of delirium: Pre-Interventional Preventive Risk Assessment (PIPRA) Tool. The importance of assessing the risk for post-operative delirium (POD) includes: providing clinicians and patients with accurate predictive information regarding the patient's risk for developing delirium as part of the risk/benefit calculation for surgical procedures, and thus potential risk of subsequent cognitive impairment; as well as the ability to introduce timely prophylactic techniques that may prevent its onset.

The PIPRA tools consists of nine items commonly found in any presurgical patient's electronic medical record (EMR). The tool has been designed to run in the background of the EMR and automatically calculate the patient's risk for developing delirium upon admission for surgical intervention. For our study, we will be applying the PIPRA tool to the EMR of patients already enrolled in a parallel study as detailed above.

The PIPRA tool predicts the risk of developing POD delirium based on its algorithm that takes into consideration the following nine clinical variables: age, height/weight or body mass index, the American Society of Anesthesiologist physical status Classification system (ASA), past history of delirium, past history of cognitive impairment (including dementia), number of medications, preoperative C-reactive protein levels, surgical risk (as determined by the European Society of Anesthesiology), and type of surgery. The subsequent result predicts the risk (in percentage) of a patient developing POD following surgery.

The PIPRA tool is fully integrated into EMR systems, operating in the background, extracting relevant information, and automatically generating a delirium prediction score. In addition, this software possesses the flexibility to recalibrate the delirium risk based on the availability of the nine clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients
* Greater than or equal to 65 years old
* ASA I, II or III
* Greater than 90 min of surgery
* Non-cardiac surgery

Exclusion Criteria:

* Dementia
* Alzheimer's
* Parkinson's
* Current Benzodiazepine use
* Alcoholism
* Previous surgery within the last 12 months or expected in the 12 months to come (except the expected surgery for which they are being enrolled).
* Color-blindness

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Stanford Hospital geriatric patients having surgery
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with postoperative delirium accurately predicted by the PIPRA Tool | Baseline measurement of variables and detection of delirium presenting up to 72 hours post-operatively
  Assessment of the accuracy on the prediction of subjects identified as developing delirium by the PIPRA tool, as compared with post-operative standardized delirium assessment tools. We will compare the assessment of the PIPRA prediction tool (performed pre-op) with the actual development of delirium as assessed by a clinical assessment based on DSM; the CAM-ICU & SPTD assessment tools.
Development of post-operative Delirium | Up to 72 hours post-operatively
  Number of subjects diagnosed with post-operative delirium
Determination of Delirium Phenotype | Up to 72 hours post-operatively.
  For those who develop delirium, the phenotype of delirium will be determined as per the Liptzin-Levkoff Criteria (based on DSM diagnostic Criteria). As such, all delirium episodes will be categorized as: hyperactive, hypoactive, mixed, or subsyndromal delirium.
Impact of delirium on post-operative cognitive impairment | Up to 10-year post-operatively.
  Impact of delirium occurrence and emergence of cognitive impairment post-operatively
Sensitivity and specificity of the PIPRA tool for detecting postoperative delirium. | Baseline measurement of variables and detection of delirium presenting up to 72 hours post-operatively
  Sensitivity and specificity of various cut off points of the PIPRA tool for detecting postoperative delirium.
Receiver operating characteristic (ROC) curve analysis of PIPRA tool | Baseline measurement of variables and detection of delirium presenting up to 72 hours post-operatively
  Receiver operating characteristic (ROC) curve analysis of PIPRA tool

SECONDARY OUTCOMES:
Immediate Postoperative Mortality | From date of post-operative admission up to time of postoperative discharge, an average of 72 hours.
  Mortality rate immediately after index surgery
Length of Hospital Length of Stay | From date of post-operative admission up to time of postoperative discharge (assessed up to 1 year after admission).
  Total number of days admitted to the hospital
Discharge Site | Type of facility the patient was discharge to from the hospital (assessed up to 6 months from admission)
  Site of discharge (e.g., home, rehabilitation, skilled nurse facility, etc)
Requirement of Intensive Care Unit Admission | Time to discharge from the hospital (assessed up to 6 months from admission)
  Need for admission to an intensive care unit due to clinical necessity or deterioration
Need of pharmacological protocol | From post-operative hospital admission up to time of postoperative discharge (assessed up to 6 months from admission)
  Need of pharmacological protocol for management of delirium

CONTACTS AND LOCATIONS:
Overall Officials: José R Maldonado, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medical Center, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buchan TA, Sadeghirad B, Schmutz N, Goettel N, Foroutan F, Couban R, Mbuagbaw L, Dodsworth BT. Preoperative prognostic factors associated with postoperative delirium in older people undergoing surgery: protocol for a systematic review and individual patient data meta-analysis. Syst Rev. 2020 Nov 14;9(1):261. doi: 10.1186/s13643-020-01518-z. PMID 33189147
- [Result] Dodsworth BT, Reeve K, Falco L, Hueting T, Sadeghirad B, Mbuagbaw L, Goettel N, Schmutz Gelsomino N. Development and validation of an international preoperative risk assessment model for postoperative delirium. Age Ageing. 2023 Jun 1;52(6):afad086. doi: 10.1093/ageing/afad086. PMID 37290122
- [Result] Sadeghirad B, Dodsworth BT, Schmutz Gelsomino N, Goettel N, Spence J, Buchan TA, Crandon HN, Baneshi MR, Pol RA, Brattinga B, Park UJ, Terashima M, Banning LBD, Van Leeuwen BL, Neerland BE, Chuan A, Martinez FT, Van Vugt JLA, Rampersaud YR, Hatakeyama S, Di Stasio E, Milisen K, Van Grootven B, van der Laan L, Thomson Mangnall L, Goodlin SJ, Lungeanu D, Denhaerynck K, Dhakharia V, Sampson EL, Zywiel MG, Falco L, Nguyen AV, Moss SJ, Krewulak KD, Jaworska N, Plotnikoff K, Kotteduwa-Jayawarden S, Sandarage R, Busse JW, Mbuagbaw L. Perioperative Factors Associated With Postoperative Delirium in Patients Undergoing Noncardiac Surgery: An Individual Patient Data Meta-Analysis. JAMA Netw Open. 2023 Oct 2;6(10):e2337239. doi: 10.1001/jamanetworkopen.2023.37239. PMID 37819663
- [Result] Maldonado JR. Acute Brain Failure: Pathophysiology, Diagnosis, Management, and Sequelae of Delirium. Crit Care Clin. 2017 Jul;33(3):461-519. doi: 10.1016/j.ccc.2017.03.013. PMID 28601132
- [Result] Robinson TN, Eiseman B. Postoperative delirium in the elderly: diagnosis and management. Clin Interv Aging. 2008;3(2):351-5. doi: 10.2147/cia.s2759. PMID 18686756